CLINICAL TRIAL: NCT05822765
Title: Effect of Adrenaline Concentration in Tumescence Solution on Intraoperative Hemodynamics of Liposuction Patients: A Randomized Controlled Trial
Brief Title: Effect of Adrenaline Concentration on Intraoperative Hemodynamics of Liposuction Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Collaborators: Benha University (Other)
Responsible Party: Principal Investigator, Neveen Abd El Maksoad Kohaf, Lecturer of Clinical Pharmacy, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RC.3.1.2023
Record Dates: First submitted 2023-04-10; First posted 2023-04-21 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Intraoperative Hemodynamics; Liposuction
Keywords: Adrenaline; Tumescence Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Tumescence fluid contained Epinephrine concentration of 1:1000000 (one ampoule 1 mg per liter) Llidocaine 500 mg and sodium bicarbonate 8.4% 10 ml per liter.
  Interventions: Drug: Epinephrine concentration of 1:1000000
- Group B (Active Comparator): Tumescence fluid contained Epinephrine concentration of 1:500000 two ampoule 2 mg/liter.
  Lidocaine 500 mg and sodium bicarbonate 8.4% 10 ml per liter.
  Interventions: Drug: Epinephrine concentration of 1:500000

INTERVENTIONS:
Drug: Epinephrine concentration of 1:1000000 — Tumescence fluid contained Epinephrine concentration of 1:1000000 (one ampoule 1 mg per liter) lidocaine 500 mg and sodium bicarbonate 8.4% 10 ml per liter
  Arms: Group A
Drug: Epinephrine concentration of 1:500000 — Tumescence fluid contained Epinephrine concentration of 1:500000 two ampoule 2 mg/liter with same lidocaine and bicarbonate dose. lidocaine 500 mg and sodium bicarbonate 8.4% 10 ml per liter
  Arms: Group B

SUMMARY:
Liposuction is a procedure that has emerged over the last 30 years as a method to remove subcutaneous fat for cosmetic purposes. Numerous liposuction techniques have been developed .Tumescent liposuction involves using large volumes of dilute local anesthetic and epinephrine to facilitate anesthesia and decrease blood loss. Questions remain about the appropriate dose of local anesthetic, the use of general anesthesia in liposuction, and the setting in which the chosen liposuction method is used. Adrenaline is the most commonly used vasoconstrictor, the recommended concentration in the tumescent solution is 0.25-1 mg/L depending on the tissue vascularity. In the more vascular tissues, the concentration is 1 mg/L and is decreased to 0.5 mg/L in the less vascular areas of the body. The dose should not exceed 50μg/kg. If the maximum dose is anticipated to exceed, the procedure should be done in several stages.

ELIGIBILITY:
Inclusion Criteria:

* ASA I patients
* scheduled for liposuction for abdomen and flanks and body contouring with liposuction

Exclusion Criteria:

* Bleeding disorders, anemia or hemoglobin level less than 11g/dl
* Cardiovascular diseases,
* Uncontrolled diabetes mellitus,
* Collagen disorders, and
* Pregnancy

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 4 hours
  Noninvasive Blood pressure will be recorded

SECONDARY OUTCOMES:
Heart rate | 4 hours
  Heart rate will be recorded every 10 minutes and results will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Neveen Kohaf, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
data can be shared upon reasonable request from the corresponding author
Supporting Information: Study Protocol, SAP